CLINICAL TRIAL: NCT04162015
Title: Feasibility and Safety of Neoadjuvant Nivolumab and Chemotherapy for Resectable Malignant Pleural Mesothelioma
Brief Title: A Study of Nivolumab and Chemotherapy Followed by Surgery for Mesothelioma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-272
Record Dates: First submitted 2019-11-12; First posted 2019-11-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Nivolumab; Surgery; Pemetrexed; Cisplatin; Carboplatin; 19-272
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Nivolumab; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: This is a single institution pilot study of nivolumab with pemetrexed and cisplatin or carboplatin prior to surgery for patients with potentially resectable malignant pleural mesothelioma (MPM).
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- nivolumab with pemetrexed and cisplatin or carboplatin (Experimental): Eligible patients will receive two cycles of neoadjuvant therapy with nivolumab 360 mg, pemetrexed 500 mg/m2, and cisplatin 75 mg/m2 or carboplatin AUC=5. Subsequently, they will undergo pleurectomy/decortication.
  Interventions: Drug: Nivolumab; Drug: Pemetrexed; Drug: Cisplatin or Carboplatin

INTERVENTIONS:
Drug: Nivolumab — nivolumab 360 mg
Drug: Pemetrexed — 500 mg/m^2
Drug: Cisplatin or Carboplatin — cisplatin 75 mg/m2 or carboplatin AUC=5

SUMMARY:
This study will test whether giving nivolumab in combination with pemetrexed and either cisplatin or carboplatin before surgery is a safe and effective approach to treating resectable mesothelioma without delaying surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Karnofsky performance status > 70%
* Pathologic diagnosis of malignant pleural mesothelioma.
* Potentially resectable by pleurectomy/decortication, as assessed by thoracic surgeon
* Negative serum pregnancy test in women of childbearing potential
* Female patients of childbearing potential must agree to use a highly effective form of contraception for the duration of the study and for at least 5 months after the last administration of nivolumab and at least 6 months after last administration of pemetrexed, whichever is longer
* Male patients with female partners of childbearing potential must agree to use a highly effective form of contraception for the duration of the study and for at least 7 months after the last administration of nivolumab and at least 3 months after the last administration of pemetrexed, whichever is longer
* Adequate archival or fresh tissue for correlative analysis. Archival tissue will be deemed acceptable as long as their was no interval therapy prior to cycle 1 day 1 of protocol therapy. If sufficient archival or fresh tissue is not available, then a repeat biopsy at baseline prior to starting study treatment will be required as long as medically safe and feasible
* Absolute neutrophil count ≥ 1000/mcL
* Total bilirubin ≤ 1.5 mg/dl
* AST and ALT ≤ 3.0 x upper limit of normal
* Creatinine ≤ 1.5 x upper limit of normal
* Negative HIV serology blood test

Exclusion Criteria:

* Prior treatment with chemotherapy or immunotherapy for mesothelioma
* Autoimmune disease requiring systemic immune modulating treatment during the past two years
* Pregnant or lactating women
* Known active hepatitis B or hepatitis C
* Current use of systemic prednisone at dose ≥ 10 mg daily (or the equivalent dose with another corticosteroid)
* Serious concurrent medical illness or another active cancer requiring treatment
* Active pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
number of patients going to operating room for surgical resection | 30 days of the initially planned date
  Patients who experience a greater than 30 day toxicity induced delay of surgery will be counted as a failure for the primary feasibility endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Offin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memoiral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm